CLINICAL TRIAL: NCT00845091
Title: Cardiac Autonomic Regulation Enhancement Through Exercise Trial
Acronym: CARE-E
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The Miriam Hospital (Other)
Responsible Party: Principal Investigator, Eva R. Serber, Assistant Professor (Research), The Miriam Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HL092340; R21HL092340-01A1 (NIH); RIH IRB, CMTT: 0177-08
Record Dates: First submitted 2009-02-13; First posted 2009-02-16 (Estimated); Last update posted 2014-01-08 (Estimated); Status verified 2014-01

CONDITIONS: Cardiovascular Disease, Arrhythmias
Keywords: Parasympathetic activity; Exercise; Education; Arrhythmias; Defibrillators, Implantable
MeSH Terms: conditions — Cardiovascular Diseases; Arrhythmias, Cardiac; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Exercise (Experimental): moderate-intensity, low-impact, supervised, aerobic exercise
  Interventions: Behavioral: Exercise
- Heart Healthy Education (Active Comparator): Educational topics on heart health (e.g., nutrition, smoking, sleep)
  Interventions: Behavioral: Heart Healthy Education

INTERVENTIONS:
Behavioral: Exercise — moderate-intensity, low-impact, supervised, aerobic exercise
  Arms: Exercise
Behavioral: Heart Healthy Education — Educational topics related to heart health (e.g., nutrition, smoking, sleep)
  Arms: Heart Healthy Education

SUMMARY:
The current research study proposes to examine participants with implantable cardioverter defibrillators (ICD) who are randomly assigned to either an exercise training program intervention or a heart healthy education program intervention. We will look at changes in the functioning of the autonomic nervous system over time and between intervention groups. We are also going to be looking at changes in frequencies of the ICD participants' heart arrhythmias and ICD therapies (e.g., pacing, shock).; as well as, changes in exercise tolerance, psychological well-being, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* adult ICD patients (≥ 18 years of age)
* received an ICD for secondary prevention, cardiac diagnosis of: ventricular fibrillation, OR ventricular tachycardia, OR cardiac arrest, OR syncope with ventricular tachycardia inducible by programmed stimulation (EPS), AND
* either diagnosed coronary artery disease AND/OR prior myocardial infarction, or non-ischemic dilated cardiomyopathy
* meet functional NYHA Class I or II heart failure or angina symptoms
* ICD patients need to be sedentary, defined as not engaging in structured exercise more than once weekly, or an accumulation of less than 60 minutes of moderate intensity aerobic activity over the course of the week, for the past 3 months.
* deemed medically stable by their cardiologist and have received approval by their cardiologist to engage in an exercise program
* Stable (unchanged) cardiac and psychopharmacologic medications in the 3 months prior to study enrollment
* Able to read and write English
* able to commit to the 3-month exercise/heart healthy program attending 3 times per week (36 sessions)
* able to commit to the 3 assessments (pre, post-treatment, 3-month follow-up; 6-month duration)

Exclusion Criteria:

* Patients who meet functional NYHA Class III or IV heart failure or angina symptoms
* sinus node dysfunction that requires atrial pacing
* atrial fibrillation
* bi-ventricular ICD
* are pacemaker-dependent
* diagnosis of Brugada's Syndrome
* diagnosis of arrhythmogenic right ventricular dysplasia
* complex congenital heart disease
* orthopedic restrictions, limitations, or disabilities that would jeopardize the patient's safety during exercise or form completing the treadmill stress test
* Neurocognitive or cognitive impairments that will result in nonadherence (based on clinical evaluation)
* Unstable angina
* resting systolic blood pressure >180mmHg or resting diastolic blood pressure >110mm Hg will be evaluated on a case-by-case basis
* orthostatic blood pressure drop of >20mm Hg with symptoms
* critical aortic stenosis (peak systolic pressure gradient >50mm Hg with aortic valve orifice area <0.75cm2 in average size adult)
* acute systemic illness or fever
* uncontrolled atrial or ventricular arrhythmias
* uncontrolled sinus tachycardia (>120 beats/min)
* uncompensated CHF
* 3rd degree AV block (without pacemaker)
* active pericarditis or myocarditis
* recent embolism; thrombophlebitis
* resting ST segment displacement (>2mm)
* uncontrolled diabetes (resting blood glucose >400mg/dl)
* metabolic problems, such as acute, hypo or hyperkalemia, hypovolemia
* recent strongly positive exercise test as achieved by: significant decrease in systolic blood pressure with increasing workload, OR early onset, horizontal or downsloping ST segment depression (4mm), OR prolonged electrocardiogram (ECG) changes during recovery
* hypertrophic obstructive cardiomyopathy
* severe pulmonary hypertension
* patients who do not pass the exercise stress test

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2009-02; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
parasympathetic activity and regulation | 3 months, 6 months

SECONDARY OUTCOMES:
arrhythmia frequency | 3 months, 6 months
ICD therapy frequency | 3 months, 6 months
exercise tolerance | 3 months, 6 months
psychological well-being | 3 months, 6 months
quality of life | 3 months, 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Eva R Serber, Ph.D., Principal Investigator — The Miriam Hospital
Locations (1):
- The Miriam Hospital Centers for Behavioral and Preventive Medicine, Providence, Rhode Island, United States

REFERENCES:
- [Background] Palmer K, Tilkemeier PL, Buxton AE, Niaura R, Marcus B, Todaro J, Serber ER. Ratings of perceived exertion and physiological responses during exercise testing among ICD patients. Poster presented at the 32nd Annual Meeting of the Society for Behavioral Medicine, New Orleans, LA.; Abstract B-1621, Rapid Communications, April 2012.